CLINICAL TRIAL: NCT00129727
Title: Phase II Evaluation of Carboplatin, Paclitaxel and Bevacizumab as First Line Chemotherapy and Consolidation for Advanced Ovarian Cancer
Brief Title: Carboplatin Taxol Avastin in Ovarian Cancer (OVCA)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Women and Infants Hospital of Rhode Island (Other)
Responsible Party: Principal Investigator, Richard Thomas Penson, Clin Dir Med Gyn Onc, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04-247
Record Dates: First submitted 2005-08-10; First posted 2005-08-12 (Estimated); Results first posted 2016-06-01 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-04

CONDITIONS: Ovarian Cancer
Keywords: Carboplatin; Paclitaxel; Bevacizumab; Ovarian; Cancer
MeSH Terms: conditions — Ovarian Neoplasms; Neoplasms | interventions — Paclitaxel; Carboplatin; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Phase II (Experimental): Paclitaxel carboplatin bevacizumab
  Interventions: Drug: Paclitaxel; Drug: Carboplatin; Drug: Bevacizumab

INTERVENTIONS:
Drug: Paclitaxel — Given intravenously
  Other Names: Taxol
Drug: Carboplatin — Given intravenously
  Other Names: CBDCA
Drug: Bevacizumab — Given intravenously
  Other Names: Avastin

SUMMARY:
Study Design: This ia a Phase II study.

Subjects: Patients with chemotherapy naive epithelial ovarian cancer; or fallopian, primary peritoneal and papillary serous mullerian tumors will be recruited.

Carboplatin and Taxol (paclitaxel) will be administered concurrently with bevacizumab after surgery for 6-8 cycles every 21 (q21) days. Bevacizumab will be omitted in the first cycle, immediately post-operatively. This will be followed by one year of bevacizumab q21.

Outcomes: Outcomes include toxicity, response rate, and progression free survival.

DETAILED DESCRIPTION:
Ovarian cancer is diagnosed in approximately 26,000 American women each year, and is the leading cause of death from gynecologic cancers. Difficult to detect, the disease typically presents only when advanced. Ovarian cancer is among the most sensitive of solid tumors to chemotherapy. However, the majority of patients with ovarian cancer who achieve a complete remission with first line platinum-based chemotherapy will ultimately develop recurrent disease. The combination of carboplatin and paclitaxel is the standard first line combination in the US.

In patients with advanced ovarian cancer, carboplatin plus paclitaxel results in less toxicity, is easier to administer, and is not inferior, when compared with cisplatin plus paclitaxel. The randomized trial, GOG-158 finally confirmed the adoption of this standard with an improved toxicity profile of the combination of cisplatin and paclitaxel, a doublet that had been previously demonstrated to have a substantially better progression free and overall survival advantage compared with cisplatin and cyclophosphamide in advanced-stage epithelial ovarian cancer. Although in nonrandomized trials, carboplatin and paclitaxel was a less toxic and highly active combination regimen, there remained concern regarding its efficacy in patients with good prognosis completely resected advanced disease.

In parallel European, multicentre, randomised trials, between January, 1996, and March, 2002, 802 patients with platinum-sensitive ovarian cancer relapsing after 6 months of being treatment-free were enrolled from 119 hospitals in five countries (ICON III). Patients were randomly assigned paclitaxel plus platinum chemotherapy or conventional platinum-based chemotherapy. Survival curves demonstrated a difference in favor of paclitaxel plus platinum (hazard ratio 0.82 [95% CI 0.69-0.97], p=0.02), corresponding to an absolute difference in 2-year survival of 7% between the paclitaxel and conventional treatment groups (57 vs 50% [95% CI for difference 1-12]), and median survival of 5 months (29 vs 24 months [1-11]).

Since the hypothesis of targeting angiogenesis to treat cancer was first described in 1971 by Judah Folkman, there has been intense research into the development of antiangiogenic cancer therapies. Tumors are dependent on their development of a vascular supply. Recent work has shown that, if cells are already transformed, angiogenesis can be initiated with a tumor mass comprising as few as 100-300 cells.

VEGF actions are mediated through binding to two receptor tyrosine kinases, VEGF-R-1 (Flt-1) and VEGF-R- 2 (KDR; whose murine form is known as Flk-1). Activation of these receptors by VEGF triggers the phosphorylation of a multitude of proteins that are active in signal transduction cascades. VEGF gene expression is upregulated by a wide range of stimuli including hypoxia, nitric oxide, estrogen, a variety of growth factors (e.g., FGF-4, PDGF, TNF, TGF-b, EGF, IL-6, IL-1b, #76) and common genetic events associated with the malignant phenotype (loss of tumor suppressor genes such as p53 and activation of oncogenes such as ras, v-src and HER2/neu). Beside major angiogenic properties, VEGF is a potent mitogen for vascular endothelium, inhibits endothelial apoptosis and mobilizes bone marrow-derived endothelial cell precursors. VEGF also mediates the secretion of enzymes involved in the degradation of extracellular matrix, modulates migration, increases vascular permeability, upregulates hexose transport and induces monocyte migration.

Ovarian cancers secrete large amounts of VEGF in vitro and in vivo, and VEGF appears to play a crucial role in angiogenesis and tumor induced immunosuppression in ovarian cancer patients. Indeed, VEGF has been confirmed as an independent prognostic indicator by multivariate analysis of survival.

Angiogenesis is crucial in the development of ovarian cancer. VEGF is closely linked to normal ovarian function and is required for the development of the corpus luteum and the maturation of the endometrium. Elevated VEGF expression occurs in all stages of ovarian cancer and is associated with poor prognosis. In fact, VEGF levels appear to be prognostically important. In addition to its role in ovarian-cancer-associated angiogenesis, VEGF overexpression is directly associated with the production of ascitic fluid, a feature probably related to its ability to induce endothelial hyperpermeability. In studies monitoring VEGF after tumor resection, VEGF appears to be a valid tumor marker, following a dramatic decline after surgery, the levels rise at recurrence.

The parent murine antibody of bevacizumab, A.4.6.1, demonstrated promising antitumor activity in a subcutaneous SKOV-3 human ovarian cancer xenograft model. Interestingly, in the intraperitoneal model of the same cell line, A.4.6.1 produced only partial inhibition of tumor growth, but was associated with almost complete inhibition of ascites production. These data provided the rationale for evaluation of bevacizumab in ovarian cancer. A Gynecologic Oncology Group (GOG) phase II study of bevacizumab monotherapy is ongoing, and a second trial will examine the combination of bevacizumab with daily, low-dose, oral cyclophosphamide, using metronomic dosing in the hope that 'less is more'.

Bevacizumab (rHumAb VEGF; Genentech, Inc., CA), a recombinant humanized monoclonal antibody directed to VEGF, and neutralizes the biological properties of human VEGF. Bevacizumab, derived from the murine antibody A.4.6.1, comprises 93% human IgG frameworks and 7% murine-derived antigen-binding regions, the humanization providing a longer half-life and less immunogenicity.

Based on preclinical data, a phase I/II program with bevacizumab was initiated. The initial phase I trial enrolled 25 patients in a dose-escalation fashion (0.1-10.0 mg/kg on days 0, 28, 35, and 42). No grade 3 or 4 toxicity was seen that was directly attributable to therapy. There were three episodes of tumor-related bleeding, including a hemorrhage in a previously undetected cerebral metastasis. Grade 1 and 2 toxicities, possibly or probably related to treatment, included asthenia, headache, and nausea. There were no complete or partial responses seen, although one patient with renal cell carcinoma achieved a mixed response.

The material use in this study is NOT commercially available Avastin™ (Genentech, Inc.; South San Francisco, CA), and may differ from that product.

Bevacizumab demonstrated preclinical and clinical activity in colorectal cancer and Genentech chose this as the disease for their registration studies. At ASCO 2003 Hurwitz et al reported the results of their phase III study of standard bolus irinotecan/5-FU/LV (IFL) plus bevacizumab (5 mg/kg). An impressive median survival advantage (20.3 months vs. 15.6 months [p=0.00003]) was reported in 925 patients receiving first line therapy with irinotecan, 5-fluorouracil, leucovorin treatment for metastatic colorectal cancer. Only grade 3 hypertension (11%), easily managed with oral medications, was clearly increased in this Phase III study. Gastrointestinal perforation, although rare, was possibly seen more frequently.

Importantly, this was the first phase III validation of an antiangiogenic approach for the treatment of human cancer. Several further, large phase III trials of bevacizumab in metastatic colorectal cancer are under way. These include a first-line study of standard 5-FU/LV with or without bevacizumab in patients who are not appropriate for irinotecan therapy. A further phase III study will assess the FOLFOX regimen with or without bevacizumab in the second-line setting for patients who have failed previous irinotecan plus 5-FU treatment. These results will help to define the benefit of anti-VEGF therapy.

Other studies are awaited, notably ECOG 4599 a randomized comparison of Taxol and carboplatin with and without bevacizumab, in patients with non-small cell lung cancer has completed accrual with over 600 patients.

There are three reasons to investigate protracted exposure to bevacizumab. Firstly, the agent, while inducing apoptosis, is considered a cytotoxic and protracted exposure is thought to be necessary to maintain tumor dormancy. Secondly, the studies in colorectal cancer treated patients until tumor progression. Lastly, there is an evolving paradigm in the treatment of ovarian cancer. It is now widely accepted that continual rather than intermittent palliative chemotherapy translates into a better quality of life. The Gynecologic Oncology Group have recently reported a provocative randomized controlled trial that confirmed a significant and large improvement in progression free survival (GOG 178), considered the most important end point in the patients with advanced ovarian cancer. Furthermore, in the preclinical studies of ovarian cancer, the ovarian cancer model presented a compelling argument for prolonged bevacizumab administration. Having inoculated the human ovarian carcinoma cell line SKOV-3 within the peritoneal cavity of immunodeficient mice, tumor engrafted in 7 to 10 days. The function-blocking VEGF antibody, A4.6.1 significantly inhibited subcutaneous SKOV-3 tumor growth approximately 20 fold compared with controls (P < 0.05), and similarly in the intraperitoneal model. Importantly, within 2 to 3 weeks of cessation of A4.6.1 treatment, effectively treated mice developed severe ascites, became cachectic, and had to be killed, and subsequent tumor burden in these animals varied from moderate to high. It should be clarified that the murine study utilized A4.6.1 the murine precursor of bevacizumab, but that the results can be extrapolated to the actions of bevacizumab.

OVERVIEW OF TRIAL DESIGN Study Design: Open label phase II study. Subjects: Patients with chemotherapy naive epithelial ovarian cancer; or fallopian, primary peritoneal and papillary serous mullerian tumors .

CHEMOTHERAPY Carboplatin and paclitaxel administered concurrently with bevacizumab after surgery for for 6-8 cycles q21 days. Bevacizumab will be omitted in the first cycle, immediately post-operatively and continued for one year of consolidation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older.
* Histological diagnosis of epithelial ovarian carcinoma, fallopian tube cancer, primary peritoneal carcinoma or papillary serous mullerian carcinoma.
* Previous attempted surgical debulking.
* Stage IC or greater.
* Performance status 0-2 by the ECOG scale.
* Peripheral neuropathy < grade 2.
* Life expectancy must be >= 6 months.
* Patients must be informed of the investigational nature of the study and sign an informed consent form.

Exclusion Criteria:

* History of serious systemic disease, including: myocardial infarction within the last 6 months; uncontrolled hypertension (blood pressure of >160/110 mmHg on medication); unstable angina; New York Heart Association (NYHA) Grade II or greater congestive heart failure; unstable symptomatic arrhythmia requiring medication (subjects with chronic atrial arrhythmia, i.e., atrial fibrillation or paroxysmal supraventricular tachycardia are eligible); or peripheral vascular disease (Grade II or greater). Prior history of thrombotic events and stroke are also included as exclusion criteria.
* Neutrophil count <1,500/mm3; platelet count <100,000/m3.
* Alkaline phosphatase or bilirubin > 1.5 x upper limit of normal (ULN); SGOT > 5 x ULN.
* Calculated creatinine clearance < 50 ml/min.
* Prior chemotherapy or radiotherapy.
* Inadequate surgical cytoreduction such that interval cytoreductive surgery could materially improve prognosis. Patients are not permitted to have interval cytoreductive surgery on study.
* Concurrent invasive malignancy. (Patients with concurrent superficial endometrioid endometrial carcinoma are eligible, if their endometrial carcinoma is superficial or invades less than 50% of the thickness of the myometrium.)
* Uncontrolled hypertension (defined as a Grade 4 event that has failed to resolve with observation or treatment) or bleeding diathesis.
* Evidence of tumor involving major blood vessels on any prior computed tomography (CT) scan.
* Surgical wound that has failed to close.
* Prior treatment with an anti-angiogenic agent.
* Any active bleeding.
* Therapeutic anticoagulation (prophylactic very low dose warfarin is allowed [1mg by mouth (p.o.) once daily (qd) with International Normalized Ratio (INR) <1.2]).
* Active psychiatric disease or neurologic symptoms requiring treatment (Grade I sensory neuropathy allowed).
* Presence of central nervous system or brain metastases.
* Proteinuria at baseline or clinically significant impairment of renal function. Subjects unexpectedly discovered to have > 1+ proteinuria at baseline should undergo a 24-hour urine collection, which must be an adequate collection and must demonstrate < 1g of protein/24 hr to allow participation in the study.
* Dementia or significantly altered mental status that would prohibit the understanding and/or giving of informed consent.
* Patients with known hypersensitivity to Cremophor EL.
* Patients with active bacterial, viral or fungal infections
* Patients receiving other investigational therapy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2005-06; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard T Penson, MRCP MD, Principal Investigator — MGH

IPD SHARING:
Plan to Share IPD: Yes
Manuscript was published in JCO

REFERENCES:
- See also: URL is the published abstract — http://www.ncbi.nlm.nih.gov/pubmed/19917843

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred during the planned time frame. Recruitment occurred at Massachusetts General Hospital; Dana-Farber Cancer Institute; Beth Israel Deaconess Medical Center; and Women and Infants Hospital of Rhode Island.
Groups:
- Phase II of Carboplatin, Pacitaxel, and Bevacizumab: Phase II Evaluation of Carboplatin, Pacitaxel, and Bevacizumab as First Line Chemotherapy and Consolidation for Advanced Ovarian Cancer.
Period: Overall Study
Arm/Group | Phase II of Carboplatin, Pacitaxel, and Bevacizumab
Started | 62
Completed | 57
Not Completed | 5

BASELINE CHARACTERISTICS:
Arm/Group | Phase II of Carboplatin, Pacitaxel, and Bevacizumab
Number analyzed (Participants) | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 44
  >=65 years | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 62

OUTCOME MEASURES:

1. Primary Outcome: PFS
Description: Progression Free Survival: To examine the toxicity, estimate the objective response rate, and progression free survival measured in months of carboplatin, paclitaxel, and bevacizumab followed by single agent bevacizumab as consolidation for advanced mullerian cancer
Time Frame: Median PFS in months - up to 5 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase II of Carboplatin, Pacitaxel, and Bevacizumab
Number analyzed (Participants) | 62
Months | 29.8 [17.3 to NA] — NA = Upper limit not yet reached

2. Secondary Outcome: Response Rate (RECIST-1)
Description: To estimate the objective response rate of carboplatin, paclitaxel, and bevacizumab. Evaluate toxicity.
Time Frame: 5 years
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Phase II of Carboplatin, Pacitaxel, and Bevacizumab
Number analyzed (Participants) | 62
Percentage of Participants | 76 [69 to 87]

3. Secondary Outcome: Toxicity
Description: Per CTCAE (Common Toxicity Criteria for Adverse Events) number of participants who experienced toxicity on the study
Time Frame: 60 months
Measure: Number; unit: Participants
Arm/Group | Phase II of Carboplatin, Pacitaxel, and Bevacizumab
Number analyzed (Participants) | 62
Participants | 62

ADVERSE EVENTS:
Time Frame: 5 years
Description: CTCAE version 3
Arm/Group | Phase II of Carboplatin, Pacitaxel, and Bevacizumab
Serious Adverse Events (participants affected / at risk) | 9/62
Other Adverse Events (participants affected / at risk) | 2/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase II of Carboplatin, Pacitaxel, and Bevacizumab (N=62)
Peripheral neuropathy (Nervous system disorders) | 1 (1)
GI perforation (Gastrointestinal disorders) | 1 (1)
Wound infection (Skin and subcutaneous tissue disorders) | 1 (1)
Pulmonary embolus (Vascular disorders) | 2 (2)
Hypotension (General disorders) | 1 (1)
nasal perforation (Musculoskeletal and connective tissue disorders) | 1 (1)
abdominal pain (General disorders) | 1 (1)
SVT (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase II of Carboplatin, Pacitaxel, and Bevacizumab (N=62)
Hem toxicty (Blood and lymphatic system disorders) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Phase II uncontrolled trial

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days